CLINICAL TRIAL: NCT02499835
Title: Pilot Trial of pTVG-HP DNA Vaccine and Pembrolizumab in Patients With Castration-Resistant, Metastatic Prostate Cancer
Brief Title: Vaccine Therapy and Pembrolizumab in Treating Patients With Hormone-Resistant, Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Prostate Cancer Foundation (Other); Madison Vaccines Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW15014; 2015-0453 (Other: IRB); NCI-2015-01154 (Registry Identifier: NCI CTRP); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 3/19/2018 (Other: UW Madison)
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Results first posted 2022-12-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Soft Tissues; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab; Immunoglobulin G

STUDY DESIGN:
Intervention Model Description: Once at least 12 subjects per arm are accrued to Arms 1 and 2, and Arm 3 is open to accrual, accrual will occur only to Arm 3 (other arms will be closed). Extended treatment Arm 4 will open only when Arm 3 has met accrual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (pTVG-HP plasmid DNA vaccine, concurrent pembrolizumab) (Experimental): Patients receive pTVG-HP plasmid DNA vaccine ID every other week on days 1, 15, 29, 43, 57, and 71 and pembrolizumab IV over 30 minutes every 3 weeks on days 1, 22, 43, and 64.
  Interventions: Biological: Pembrolizumab; Biological: pTVG-HP Plasmid DNA Vaccine
- Arm II (pTVG-HP plasmid DNA vaccine, sequential pembrolizumab) (Experimental): Patients receive pTVG-HP plasmid DNA vaccine ID as in Arm I and pembrolizumab IV over 30 minutes every 3 weeks on days 85, 106, 127, and 148.
  Interventions: Biological: Pembrolizumab; Biological: pTVG-HP Plasmid DNA Vaccine
- Extended Treatment Arm III (Experimental): pTVG-HP (100 μg) with rhGM-CSF (208 μg) administered intradermally (i.d.) every 3 weeks, for a maximum of 16 doses. Pembrolizumab 2 mg/kg, with a maximum dose of 200 mg, administered intravenously every 3 weeks, for a maximum of 16 doses, beginning on day 1 after the first pTVG-HP vaccination.
  Interventions: Biological: Pembrolizumab; Biological: pTVG-HP Plasmid DNA Vaccine
- Extended Treatment Arm IV (Experimental): pTVG-HP (100 µg) with rhGM-CSF (208 µg) administered intradermally (i.d.) every 2 weeks, for a maximum of 24 doses Pembrolizumab 2 mg/kg, with a maximum dose of 200 mg, administered intravenously every 4 weeks, for a maximum of 12 doses, beginning on day 1 after the first pTVG-HP vaccination
  Interventions: Biological: Pembrolizumab; Biological: pTVG-HP Plasmid DNA Vaccine

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: 1374853-91-4; Immunoglobulin G4; Anti-(Human Programmed Cell Death 1); Lambrolizumab; Keytruda; MK-3475; SCH 900475
Biological: pTVG-HP Plasmid DNA Vaccine — Given ID

SUMMARY:
This randomized pilot trial studies vaccine therapy and pembrolizumab in treating patients with prostate cancer that does not respond to treatment with hormones (hormone-resistant) and has spread to other places in the body (metastatic). Vaccines made from deoxyribonucleic acid (DNA), such as pTVG-HP plasmid DNA vaccine, may help the body build an effective immune response to kill tumor cells. Monoclonal antibodies, such as pembrolizumab, may find tumor cells and help kill them. Giving pTVG-HP plasmid DNA vaccine and pembrolizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of pembrolizumab in combination with pTVG-HP (pTVG-HP plasmid DNA vaccine) in patients with castration-resistant, metastatic prostate cancer.

II. To determine the 6-month progression-free survival and median time to radiographic progression in patients with castration-resistant metastatic prostate cancer treated with pembrolizumab in combination with pTVG-HP.

III. To evaluate the anti-tumor response rates (objective response rate and prostate specific antigen [PSA] response rate, using Prostate Cancer Clinical Trials Working Group 2 [PCWG2] criteria) in patients with castration-resistant metastatic prostate cancer treated with pembrolizumab in combination with pTVG-HP.

SECONDARY OBJECTIVES:

I. To determine whether either treatment sequence, or prostatic acid phosphatase (PAP)-specific immune response, is associated with prolonged (6-month) radiographic progression-free survival.

II. To evaluate effects of schedule (concurrent versus delayed administration of pembrolizumab) on the magnitude of PAP-specific T-cell responses, programmed death receptor-1 (PD-1) expression on circulating T cells, and ligands for PD-1 (PD-L1) expression on circulating epithelial cells (CEC) and on tumor biopsies.

III. To determine the median time to radiographic progression using a concurrent administration schedule

TERTIARY OBJECTIVES:

I. To evaluate effects of treatment on number of circulating tumor cells. II. To evaluate PAP-specific antibody responses following treatment with pembrolizumab and pTVG-HP DNA vaccine (pTVG-HP plasmid DNA vaccine).

III. To determine whether either treatment sequence elicits immunologic antigen spread to other prostate-associated antigens.

IV. To determine whether pre-existing or vaccine-induced PD-L1 expression on CEC or tumor biopsies is predictive of objective clinical response.

V. To determine whether treatment elicits expression of other regulatory molecules on tumor-specific T cells (e.g. hepatitis A virus cellular receptor 2 [TIM3], B and T lymphocyte associated [BTLA], and lymphocyte-activation gene 3 [LAG3]) or tumor cells (e.g. tumor necrosis factor receptor superfamily, member 14 [HVEM], phosphatidyl serine, ligands for programmed death receptor-2 [PD-2] [PD-L2]).

VI. To determine whether PD-1-regulated antigen-specific T cells identified by trans vivo delayed-type hypersensitivity (DTH) testing can identify patients who develop objective clinical responses with PD-1 blockade therapy in combination with pTVG-HP.

VII. To determine whether changes in lymph nodes and soft tissue tumor lesions are observed by fluorothymidine F-18 (FLT) positron emission tomography (PET)/computed tomography (CT) after treatment with vaccine with or without pembrolizumab.

VIII. To determine if PD-1 inhibitor therapy in combination with pTVG-HP will change number and activity (SUV) in osteoblastic metastases as measured by NaF PET/CT.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pTVG-HP plasmid DNA vaccine intradermally (ID) every other week on days 1, 15, 29, 43, 57, and 71 and pembrolizumab intravenously (IV) over 30 minutes every 3 weeks on days 1, 22, 43, and 64.

ARM II: Patients receive pTVG-HP plasmid DNA vaccine ID as in Arm I and pembrolizumab IV over 30 minutes every 3 weeks on days 85, 106, 127, and 148.

After completion of study treatment, patients are followed up 3, 6, 9, and 12 months and then annually for 2 years.

ARM III: Extended Treatment. Patients received pTVG-HP + Pembrolizumab Extended Treatment

ARM IV: Extended Treatment. Patients receive pTVG-HP every two weeks, and Pembrolizumab every 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate)
* Metastatic disease as evidenced by the presence of soft tissue and/or bone metastases on imaging studies (CT of abdomen/pelvis, bone scintigraphy)
* Castrate-resistant disease, defined as follows:

  * All patients must have received (and be receiving) standard of care androgen deprivation treatment (surgical castration versus gonadotropin-releasing hormone [GnRH] analogue or antagonist treatment); subjects receiving GnRH analogue or antagonist must continue this treatment throughout the time on this study
  * Patients may or may not have been treated previously with a nonsteroidal antiandrogen; for patients previously treated with an antiandrogen, they must be off use of anti-androgen for at least 4 weeks (for flutamide) or 6 weeks (for bicalutamide or nilutamide) prior to registration; moreover, subjects who demonstrate an anti-androgen withdrawal response, defined as a >= 25% decline in PSA within 4-6 week of stopping a nonsteroidal antiandrogen, are not eligible until the PSA rises above the nadir observed after antiandrogen withdrawal
  * Patients must have a castrate serum level of testosterone (< 50 ng/dL) within 6 weeks of day 1
* Progressive disease while receiving androgen deprivation therapy defined by any one of the following as per the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) bone scan criteria or Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 during or after completing last therapy:

  * PSA: at least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, with the final value >= 2.0 ng/mL
  * Measurable disease: >= 50% increase in the sum of the cross products of all measurable lesions or the development of new measurable lesions; the short axis of a target lymph node must be at least 15 mm by spiral CT to be considered a target lesion
  * Non-measurable (bone) disease: the appearance of two or more new areas of uptake on bone scan (or fluorine F 18 sodium fluoride [NaF] PET/CT) consistent with metastatic disease compared to previous imaging during castration therapy; the increased uptake of pre-existing lesions on bone scan will not be taken to constitute progression, and ambiguous results must be confirmed by other imaging modalities (e.g. X-ray, CT or magnetic resonance imaging [MRI])
* Prior treatment with abiraterone or enzalutamide is permitted, but patients must have been off prior corticosteroid treatment for at least 3 months
* Life expectancy of at least 6 months
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* White blood cells (WBC) >= 2000/mm^3
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Hemoglobin (HgB) >= 9.0 gm/dL
* Platelets >= 100,000/mm^3
* Creatinine =< 2.0 mg/dL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* No known history of human immunodeficiency virus (HIV) 1 and 2, human T-lymphotropic virus (HTLV)-1, or active hepatitis B or hepatitis C
* Patients must be at least 4 weeks from any prior treatments and have recovered (to < grade 2) from acute toxicity attributed to this prior treatment, unless considered chronic
* Patients must be willing and able (in the opinion of the treating physician) to undergo two research biopsies for the investigational component of this trial
* Patients must be willing to undergo two leukapheresis procedures for the investigational component of this trial
* Patients must be willing to undergo FLT PET/CT or NaF PET/CT scans for the investigational component of this trial and have no known allergies to FLT or NaF
* For those patients who are sexually active, they must be willing to use barrier contraceptive methods during the period of treatment on this trial (and for four weeks after the last DNA immunization treatment for patients in Arm 1)
* Patients must be informed of the experimental nature of the study and its potential risks, and must sign an Institutional Review Board (IRB)-approved written informed consent form indicating such an understanding

Exclusion Criteria:

* Small cell or other variant (non-adenocarcinoma) prostate cancer histology, unless there is evidence that the tumor expresses PAP
* Patients may not be receiving other investigational agents or be receiving concurrent anticancer therapy other than standard androgen deprivation therapy
* Concurrent bisphosphonate therapy is not excluded, however patients should not start bisphosphonate therapy while on this study; those patients already receiving bisphosphonate therapy should continue at the same dosing and schedule as prior to study entry
* Rapidly progressive symptomatic metastatic disease, as defined by the need for increased opioid analgesics within one month of registration for the treatment of pain attributed to a prostate cancer metastatic lesion; patients receiving opioids must receive approval from the principal investigator (PI) for eligibility
* Treatment with any of the following medications within 28 days of registration, or while on study, is prohibited:

  * Systemic corticosteroids (at doses over the equivalent of 5 mg prednisone daily) - not permitted within 3 months of registration; inhaled, intranasal or topical corticosteroids are acceptable
  * Prostate cancer (PC)-SPES
  * Saw palmetto
  * Megestrol
  * Ketoconazole
  * 5-alpha-reductase inhibitors - patients already taking 5-alpha-reductase inhibitors prior to 28 days prior to registration may stay on these agents throughout the course of therapy, but these should not be started while patients are on study
  * Diethyl stilbestrol
  * Abiraterone
  * Enzalutamide
  * Radium 223 (Xofigo)
  * Any other hormonal agent or supplement being used with the intent of cancer treatment
* External beam radiation therapy within 4 weeks of registration is prohibited, or anticipated need for radiation therapy (e.g. imminent pathological fracture or spinal cord compression) within 3 months of registration
* Major surgery within 4 weeks of registration is prohibited
* Prior cytotoxic chemotherapy (for example, but not limited to, docetaxel, mitoxantrone, cabazitaxel) within 6 months of registration is prohibited
* Patients with a history of life-threatening autoimmune disease
* Patients with a history of allergic reactions to filgrastim (GM-CSF) or the tetanus vaccine
* Patients who have undergone splenectomy
* Patients must not have other active malignancies other than non-melanoma skin cancers or superficial bladder cancer; subjects with a history of other cancers who have been adequately treated and have been recurrence-free for >= 3 years are eligible
* Patients with known brain metastases
* Any antibiotic therapy or evidence of infection within 1 week of registration
* Any other medical intervention or condition, which, in the opinion of the PI or treating physician, could compromise patient safety or adherence with the study requirements (including biopsies or leukapheresis procedures) over the primary 3-6 month treatment period
* Patients cannot have concurrent enrollment on other phase I, II, or III investigational treatment studies

NOTE: There is no exclusion for prior immune-based therapy. This includes patients previously treated on Arms 1 or 2 who are otherwise eligible for treatment on Arm 3 or 4.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G McNeel, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] McNeel DG, Eickhoff JC, Wargowski E, Zahm C, Staab MJ, Straus J, Liu G. Concurrent, but not sequential, PD-1 blockade with a DNA vaccine elicits anti-tumor responses in patients with metastatic, castration-resistant prostate cancer. Oncotarget. 2018 May 22;9(39):25586-25596. doi: 10.18632/oncotarget.25387. eCollection 2018 May 22. PMID 29876010
- [Result] McNeel DG, Eickhoff JC, Wargowski E, Johnson LE, Kyriakopoulos CE, Emamekhoo H, Lang JM, Brennan MJ, Liu G. Phase 2 trial of T-cell activation using MVI-816 and pembrolizumab in patients with metastatic, castration-resistant prostate cancer (mCRPC). J Immunother Cancer. 2022 Mar;10(3):e004198. doi: 10.1136/jitc-2021-004198. PMID 35277461
- [Derived] Scarpelli M, Zahm C, Perlman S, McNeel DG, Jeraj R, Liu G. FLT PET/CT imaging of metastatic prostate cancer patients treated with pTVG-HP DNA vaccine and pembrolizumab. J Immunother Cancer. 2019 Jan 30;7(1):23. doi: 10.1186/s40425-019-0516-1. PMID 30700328
- See also: Clinical Trials at the University of Wisconsin Carbone Cancer Center — http://www.uwhealth.org/uw-carbone-cancer-center/clinical-trials/cancer-clinical-trials/36729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from UW Hospital and Clinics from July 2015 to September 2020
Period: Overall Study
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV
Started | 13 | 13 | 20 | 20
Completed | 10 | 9 | 2 | 4
Not Completed | 3 | 4 | 18 | 16
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 18 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Disease progression | 2 | 1 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV | Total
Number analyzed (Participants) | 13 | 13 | 20 | 20 | 66
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 0 | 0 | 1 | 0 | 1
  50-59 years | 0 | 3 | 0 | 4 | 7
  60-69 years | 7 | 1 | 8 | 8 | 24
  70-79 years | 5 | 6 | 11 | 7 | 29
  80-89 years | 1 | 3 | 0 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 13 | 20 | 20 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 12 | 20 | 20 | 65
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 13 | 13 | 20 | 19 | 65
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 20 | 20 | 66

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events, Using the National Cancer Common Terminology Criteria, Version 4
Description: Toxicities will be summarized by type, as reported in the adverse events section, and total events calculated per arm.
Time Frame: Up to 23 months (Up to 12 months after completion of study treatment)
Measure: Number; unit: Adverse events
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV
Number analyzed (Participants) | 13 | 13 | 20 | 20
Adverse events | 117 | 173 | 163 | 225

2. Primary Outcome: 6-month Progression Free Survival Rate
Description: 6-month progression-free survival rate will be reported for each arm, and for overall combined study. Progression is at least a 20% increase in the sum of diameters of target lesions and a 0.5cm minimum increase, or the appearance of one or more new lesions. In order to evaluate the 6-month progression-free rate as a function of baseline time point (pretreatment or 3-months post treatment), analysis will be conducted using two different baseline values: date of randomization, and 3-months disease assessment. Central tendency is appropriate due to 20% increase and measurements being a mean of growth across time periods.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percent probability
Groups:
- Overall Combined Study: Combination of results from all 4 arms of the study
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV | Overall Combined Study
Number analyzed (Participants) | 13 | 13 | 20 | 20 | 66
percent probability | 31 [4 to 58] | 45 [16 to 74] | 44 [1 to 87] | 62 [37 to 87] | 47 [23 to 63]

3. Primary Outcome: Median Time to Radiographic Progression
Description: Median time to radiographic progression will be estimated for each, and for both study arms combined, using Kaplan-Meier method. Log-rank test will be used to perform comparison of time to radiographic progression between study arms. A one-sided 0.10 significance level will be used to conduct the comparison of the 6-month progression-free survival rate and time to radiographic progression between study arms. In order to evaluate the median time to radiographic progression as a function of baseline time point (pretreatment or 3-months post treatment), analysis will be conducted.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV | Overall Combined Study
Number analyzed (Participants) | 13 | 13 | 20 | 20 | 66
months | 5.3 [2.6 to 5.4] | 5.6 [5.0 to 11.3] | 5.6 [4.6 to 12] | 8.1 [5.3 to 10.8] | 5.6 [5.4 to 10.8]

4. Primary Outcome: Number of Participants Who Have an Objective Response
Description: Will be calculated for each study arm and for all arms combined. Complete response is the disappearance of all target lesions. Partial response is at least 30% decrease in the sum of diameters of target lesions.
Time Frame: Up to 2 years
Population: Only 25 of the 66 participants had measurable disease. These numbers reflect the number of participants with measurable disease per arm, and the number reported below reflect how many participants with measurable disease had an objective response rate.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Combined: Combination of results from all 4 arms of the study
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV | Overall Study Combined
Number analyzed (Participants) | 6 | 3 | 11 | 5 | 25
Participants | 0 | 0 | 1 | 0 | 1

5. Primary Outcome: Number of Participants Who Have a PSA Response
Description: Will be calculated for each study arm and for all arms combined. PSA complete response is a decrease in PSA to ,0.2 ng/mL; partial response is greater than or equal to 50% reduction in baseline PSA.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV | Overall Combined Study
Number analyzed (Participants) | 13 | 13 | 20 | 20 | 66
Participants
  Any PSA decline | 8 | 1 | 6 | 8 | 23
  PSA decline >50% | 2 | 0 | 2 | 2 | 6

6. Secondary Outcome: PAP-specific Immune Response
Description: Number of PAP-specific immune responses will be summarized in tabular format for each study arm and all study arms combined. A significant antigen-specific response resulting from immunization will be defined as a PAP specific response.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV | Overall Combined Study
Number analyzed (Participants) | 13 | 13 | 20 | 20 | 66
Participants | 4 | 5 | 2 | 6 | 17

7. Secondary Outcome: PAP-specific T-cell Response
Description: Number and frequencies of PAP-specific T-cell responses will be summarized in tabular format.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV
Number analyzed (Participants) | 13 | 13 | 20 | 20
Participants | 4 | 5 | 2 | 6

8. Secondary Outcome: PD-1 Expression
Description: PD-1 and PD-L1 expression levels will be summarized in terms of means, standard deviations and ranges for each study arm separately and for both arms combined. A linear regression model or a negative binomial regression model will be utilized to evaluate effects of schedule (concurrent versus delayed administration pembrolizumab) on PD-1 expression on number of circulating T cells, and PD-L1 expression on number of circulating epithelial cells. Choice of the model will be dependent on distribution of outcome variables (number of circulating T-cells and number of circulating epithelial cells).
Time Frame: Up to day 85
Population: Data was not collected because of insufficient sample size; therefore, this analysis was not performed
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: PD-L1 Expression
Description: as for outcome 8
Time Frame: Up to day 85
Population: Data was not collected due to insufficient sample size; therefoe, this analysis was not performed
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of informed consent up to 23 months.
Arm/Group | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) | Extended Treatment Arm III | Extended Treatment Arm IV
All-Cause Mortality (participants affected / at risk) | 13/13 | 9/13 | 16/20 | 9/20
Serious Adverse Events (participants affected / at risk) | 1/13 | 7/13 | 4/20 | 3/20
Other Adverse Events (participants affected / at risk) | 12/13 | 13/13 | 19/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) (N=13) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) (N=13) | Extended Treatment Arm III (N=20) | Extended Treatment Arm IV (N=20)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (pTVG-HP Plasmid DNA Vaccine, Concurrent Pembrolizumab) (N=13) | Arm II (pTVG-HP Plasmid DNA Vaccine, Sequential Pembrolizumab) (N=13) | Extended Treatment Arm III (N=20) | Extended Treatment Arm IV (N=20)
Fatigue (General disorders) | 6 (7) | 6 (8) | 0 (0) | 12 (16)
Injection site reaction (General disorders) | 5 (20) | 2 (3) | 0 (0) | 4 (18)
Chills (General disorders) | 3 (3) | 1 (3) | 0 (0) | 5 (8)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 5 (8) | 5 (8) | 18 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (6) | 4 (5) | 15 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 6 (7) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3) | 3 (4) | 8 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 8 (10)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 1 (1) | 6 (7)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 5 (10) | 7 (11) | 18 (28)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (5) | 16 (18)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2) | 5 (5) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 7 (7)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (4) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (5) | 4 (7)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 8 (8) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 2 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 5 (6) | 3 (3) | 0 (0) | 5 (8)
Hypothyroidism (Endocrine disorders) | 5 (6) | 3 (3) | 0 (0) | 4 (4)
Endocrine disorders - Other, specify (Endocrine disorders) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0) | 3 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (9) | 2 (2) | 0 (0) | 5 (5)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 2 (4) | 0 (0) | 2 (2)
Weight loss (Investigations) | 2 (3) | 1 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (4) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (7)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (6) | 0 (0) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT02499835/Prot_SAP_000.pdf